CLINICAL TRIAL: NCT01365559
Title: A Phase I/II Study of Carfilzomib as a Replacement for Multiple Myeloma Patients Failing Bortezomib-containing Regimens
Brief Title: Study of Carfilzomib for Multiple Myeloma Patients Who Are Relapsed/Refractory to Bortezomib-containing Treatments
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncotherapeutics (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IST-CAR-516
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; carfilzomib; relapsed; refractory; bortezomib; Oncotherapeutics
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Carfilzomib & Non-IMiD containing regimen (Experimental): Bortezomib is replaced with carfilzomib in a combined regimen identical to the patient's previous regimen. Regimen cannot include thalidomide or lenalidomide.
  Interventions: Drug: Group A: Carfilzomib & Non-IMiD Regimen
- Group B: Carfilzomib & IMiD containing regimen. (Experimental): Bortezomib is replaced with carfilzomib in a regimen that includes IMiDs (lenalidomide or thalidomide). Thus, the regimen is carfilzomib in an IMiD-containing regimen.
  Interventions: Drug: Group B: Carfilzomib & IMiD containing regimen.

INTERVENTIONS:
Drug: Group A: Carfilzomib & Non-IMiD Regimen — Carfilzomib will be administered intravenously starting at a dose of 20 mg/m^2 over 30 minutes for the first cycle and will then be increased to 27, 36 and 45 mg/m2 during cycles 2-4, respectively. Doses will be administered IV once daily on days 1, 2, 8, 9, 15, and 16 of each cycle. Cycles will be 28 days in length.
  Combination non-IMiD drug is dosed on the identical schedule and dosage as patient was in previous bortezomib containing regimen.
  Maintenance regimen maybe administered if patient does not progress while on study.
  Arms: Group A: Carfilzomib & Non-IMiD containing regimen
Drug: Group B: Carfilzomib & IMiD containing regimen. — Carfilzomib will be administered intravenously starting at a dose of 20 mg/m^2 over 30 minutes for the first cycle and will then be increased to 27, 36 and 45 mg/m2 during cycles 2-4, respectively. Doses will be administered IV once daily on days 1, 2, 8, 9, 15, and 16 of each cycle. Cycles will be 28 days in length.
  Combination IMiD drug is dosed on the identical schedule and dosage as patient was in previous bortezomib containing regimen.
  Maintenance regimen maybe administered if patient does not progress while on study.
  Arms: Group B: Carfilzomib & IMiD containing regimen.

SUMMARY:
This is a phase I/II multicenter, open label, nonrandomized study for patients with Multiple Myeloma (MM) who will receive treatment with carfilzomib in place of bortezomib using the same bortezomib-containing combination regimen to which a MM patient has progressed while receiving. This study will enroll 45 patients total. These patients will be resistant to bortezomib as demonstrated by progressive disease while on bortezomib or have relapsed within 12 weeks of the last dose of bortezomib in a combination regimen. Patients will be sub-divided into 2 groups in this study, treatments containing (Group A) or not containing immunomodulatory drugs (IMiDs) (Group B). Thirty patient will be enrolled into Group A and 15 patients into Group B for a total of 45 patients. Patients must have received 4 doses of a minimum of 1.0 mg/m^2 of bortezomib in no more than 4 weeks per cycle. Patients must have received at least one cycle meeting this definition and have shown progressive disease to be considered eligible. Patients who have been refractory to or relapsed within 12 weeks of the last dose of bortezomib in their most recent bortezomib-containing regimen that does not include either thalidomide or lenalidomide are eligible regardless of when patients received that regimen, as long as they meet the above criteria.

Carfilzomib will subsequently replace bortezomib using the patient's most recent bortezomib-containing regimen to which the patient progressed while receiving. Patients will be eligible if they progressed from bortezomib with an alkylating agent (melphalan or cyclophosphamide), an anthracycline (doxorubicin or pegylated liposomal doxorubicin) and/or a glucocorticosteroid (prednisone, dexamethasone or medrol)and IMiD (thalidomide or lenalidomide). The study will consist of a screening period, followed by up to eight open label treatment cycles, a final assessment to occur 28 days after the end of the last treatment cycle, a follow-up period and maintenance cycles of single agent carfilzomib.

Patient who complete the combination treatment period without progressive disease will be eligible for maintenance therapy with single-agent carfilzomib. During maintenance therapy carfilzomib will be administered at the same dose given during the last cycle of combination treatment.

ELIGIBILITY:
Inclusion:

Disease-related:

1. Have a diagnosis of MM based on standard criteria
2. Currently has MM with measurable disease, defined as a monoclonal immunoglobulin spike on serum electrophoresis of at least 0.5 gm/dL and/or urine monoclonal immunoglobulin amount of at least 200 mg/24 hours.
3. Have relapsed within 12 weeks of receiving or is refractory to their most recent bortezomib-containing regimen as long as they meet the following criteria:

   * Progressed from bortezomib-containing regimen either as a single agent or in combination with an alkylating agent (melphalan or cyclophosphamide), an anthracycline (doxorubicin or pegylated liposomal doxorubicin), IMiDs (thalidomide or lenalidomide), and/or a glucocorticosteroid (prednisone, dexamethasone or medrol)
   * Bortezomib must have been administered at 4 doses of a minimum of 1.0 mg/m2 in no more than 28 days per cycle. Subjects must have received at least one cycle meeting this definition and have shown progressive disease to be considered eligible.
   * Subject who have been refractory to their most recent bortezomib-containing regimen are eligible regardless of when the subject received that regimen, as long as they meet the above criteria and have been off the treatment for > 3 weeks.

   Definition of refractory disease: patients who meet criteria for progressive disease while currently receiving treatment.

   Demographics:
4. Age ≥ 18 years
5. Life expectancy ≥ 3 months
6. ECOG performance status 0-2 at study entry

   Laboratory tests (within 14 days prior to drug dosing on Cycle 1, Day 1)
7. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; if the bone marrow is extensively infiltrated (> 70% plasma cells) then 1.0 x 109/L
8. Hemoglobin ≥ 8 g/dL (subjects may be receiving red blood cell [RBC] transfusions in accordance with institutional guidelines)
9. Platelet count ≥ 75 × 109/L; if the bone marrow is extensively infiltrated (> 70% plasma cells) then 50 x 10^9/L
10. Creatinine clearance (CrCl) ≥ 30 mL/minute either measured or calculated. Subject with a creatinine > 15mL/min and < 30 mL/min due to significant myelomatous involvement of the kidneys may be enrolled in the study after receipt of approval from Oncotherapeutics.
11. Adequate hepatic function, with AST (SGOT) and ALT (SGPT) 3 x upper limit of normal (ULN) or 5 x ULN if hepatic metastases are present and serum total bilirubin ≤ 1.5 x ULN
12. Serum potassium > 3 and < 5

    Ethical/Other
13. Written informed consent in accordance with federal, local, and institutional guidelines.
14. Females of childbearing potential (FCBP) must agree to ongoing pregnancy testing and to practice contraception.
15. Male subjects must agree to practice contraception.

Exclusion:

Disease-related

1. Plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes (POEMS) syndrome
2. Plasma cell leukemia
3. Severe hypercalcemia, i.e., serum calcium 12 mg/dL (3.0 mmol/L) corrected for albumin
4. Received the following prior therapy:

   * Chemotherapy within 21 days of enrollment (6 wks for nitrosoureas)
   * Corticosteroids (>10 mg/day prednisone or equivalent) within 21 days of enrollment
   * Immunotherapy or antibody therapy as well as thalidomide, lenalidomide, arsenic trioxide, or bortezomib within 21 days before enrollment
   * Radiation therapy within 21 days before enrollment, receipt of localized radiation therapy does not preclude enrollment
   * Use of any other experimental drug or therapy within 28 days of enrollment

   Concurrent Conditions
5. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

   * Unstable angina or myocardial infarction within 4 months prior to enrollment
   * NYHA Class III or IV heart failure
   * Uncontrolled angina
   * Clinically significant pericardial disease
   * Severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
6. Pregnant or lactating females
7. Major surgery within 28 days prior to enrollment or has not recovered from side effects of such therapy (Kyphoplasty is not considered to be a major surgical procedure; however, the investigator is to discuss enrollment of a patient with a recent history of kyphoplasty with Oncotherapeutics).
8. Acute active infection requiring treatment with systemic antibiotics, antivirals, or antifungals within 14 days prior to receiving first dose of study drug
9. Known human immunodeficiency virus infection; baseline testing is not required
10. Active hepatitis B or C infection; baseline testing is not required
11. Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment
12. Nonhematologic malignancy within the past 5 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
13. Concurrent use of other anti-cancer agents or treatments
14. Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to enrollment
15. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib)
16. Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to enrollment
17. Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-05-02 (Actual); Primary Completion 2014-06-13 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Establish MTD, determine DLT and to determine the efficacy as assessed by the overall response rate. | Montly
  Phase I:
  • To establish the maximum tolerated dose (MTD) and determine the dose limiting toxicities (DLT) following treatment.
  Phase II:
  • To determine the efficacy as assessed by the overall response rate [CR + VGPR + PR + MR] and the Time to Progression (TTP) of disease.

SECONDARY OUTCOMES:
To establish safety and efficacy following treatment. | Montly
  Phase I:
  Obtain preliminary evidence of efficacy following treatment based on:
  * SPEP, UPEP and quantification of serum immunoglobulins
  * Bone marrow aspirates & biopsies
  * B2M
  * A roentgenographic skeletal survey of bones
  Phase II:
  Establish the safety & tolerability following treatment based on:
  * Adverse events
  * Clinical lab tests
  * Vital signs
  * Medical history & body weight measurements
  * ECOG performance status
  * Concomitant medication usage
  Both phases:
  Progression Free Survival among patients who continue onto maintenance treatment

CONTACTS AND LOCATIONS:
Overall Officials: James R Berenson, MD, Principal Investigator — James R. Berenson, MD., Inc.
Locations (9):
- United States (9):
  - Pacific Oncology and Hematology, Encinitas, California
  - Pacific Cancer Care, Salinas, California
  - Central Coast Medical Oncology, Santa Maria, California
  - James R. Berenson, MD, Inc., West Hollywood, California
  - Cancer Centers of America, Zion, Illinois
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Family Cancer Center Foundation, Inc., Memphis, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia

REFERENCES:
- [Derived] Berenson JR, Hilger JD, Yellin O, Dichmann R, Patel-Donnelly D, Boccia RV, Bessudo A, Stampleman L, Gravenor D, Eshaghian S, Nassir Y, Swift RA, Vescio RA. Replacement of bortezomib with carfilzomib for multiple myeloma patients progressing from bortezomib combination therapy. Leukemia. 2014 Jul;28(7):1529-36. doi: 10.1038/leu.2014.27. Epub 2014 Jan 16. PMID 24429497